CLINICAL TRIAL: NCT03397329
Title: A Phase 1, Randomized, Open-Label, Two-Period Crossover Study Evaluating the Relative Bioavailability and Safety of the AG-348 Tablet and Capsule Formulations After Single-Dose Administration in Healthy Adults
Brief Title: Study to Evaluate the Relative Bioavailability and Safety of the AG-348 Tablet and Capsule Formulations in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AG348-C-005
Record Dates: First submitted 2017-10-25; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence A (Active Comparator)
  Interventions: Drug: AG-348 Sequence A
- Sequence B (Active Comparator)
  Interventions: Drug: AG-348 Sequence B

INTERVENTIONS:
Drug: AG-348 Sequence A — 1. Treatment Period 1 Single 50 mg dose of AG-348 administered as a capsule formulation (2 × 25 mg capsules)
  2. Washout Period 7 days
  3. Treatment Period 2 Single 50 mg dose of AG-348 administered as a tablet formulation (1 × 50 mg tablet)
  Arms: Sequence A
Drug: AG-348 Sequence B — 1. Treatment Period 1 Single 50 mg dose of AG-348 administered as a tablet formulation (1 × 50 mg tablet)
  2. Washout Period 7 days
  3. Treatment Period 2 Single 50 mg dose of AG-348 administered as a capsule formulation (2 × 25 mg capsules)
  Arms: Sequence B

SUMMARY:
The purpose of this Phase 1, randomized, open-label, two-period crossover study is to characterize and compare the pharmacokinetic (PK) profiles and evaluate the safety of the AG-348 tablet and capsule formulations after single-dose administration in healthy adult subjects. Pharmacokinetic sampling will take place serially at specified times during conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

* Be a male or female aged 18 to 55 years, inclusive.
* Have a body mass index (BMI) of ≥ 18.5 to ≤ 29.0 kg/m2 at Screening.
* Agrees to abstain from any alcohol consumption.
* Be healthy overall with no clinically significant medical abnormalities, as determined by the Investigator through evaluation of the subject's medical history and Screening vital signs, ECG, physical examination, and laboratory assessments.

Exclusion Criteria:

* Have undergone any major surgical procedure within the 3 months prior to Screening.
* Has at Screening or has had within the 12 months prior to Screening any significant illness.
* Test positive at Screening for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), or human immunodeficiency virus (HIV).
* Have a Screening systolic blood pressure (BP) reading of ≥140 mmHg (≥150 mmHg in subjects >45 years of age) OR a diastolic BP reading of ≥90 mmHg.
* Has any history of drug or alcohol abuse within the 2 years prior to Screening.
* Is a current smoker or user of any other tobacco product.
* Have had, including by voluntary donation, > 400 mL of blood collected within the 3 months prior to Screening.
* Have taken within the 14 days prior to study drug dosing any prescription medication, over-the counter medication, or nonprescription preparation-including vitamins, minerals, phytotherapeutic/herbal/plant-derived preparations, or grapefruit juice-unless deemed acceptable by the Investigator OR have taken within the 28 days prior to study drug dosing any restricted product known to strongly induce CYP3A4 metabolism (eg, St. John's Wort).
* Have participated in another clinical research study within the 3 months prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Cmax | Pharmacokinetic sampling for AG-348 will be taken for 72 hours (3 days) after single dose
  AG-348 Maximum Plasma Concentration
AUC0-last and AUC0-∞ | Pharmacokinetic sampling for AG-348 will be taken for 72 hours (3 days) after single dose
  AG-348 Area Under the Curve

SECONDARY OUTCOMES:
Assessment of adverse events | From first dose of study drug to 10 (± 1) days after single-dose of AG-348]

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Agios Pharmaceuticals, Inc, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- Covance Clinical Research Unit, Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No